CLINICAL TRIAL: NCT05208060
Title: A Phase I/II Randomized, Prospective, Double-blind, Placebo-controlled, Single-center Study to Evaluate the Ability of Sublingual MV130 to Induce the Expression of Trained Immunity in Peripheral Blood Cells
Brief Title: Study to Evaluate the Ability of Sublingual MV130 to Induce the Expression of Trained Immunity in Peripheral Blood Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MV130-SLG-039
Record Dates: First submitted 2021-08-13; First posted 2022-01-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-09

CONDITIONS: Immune Response
Keywords: Trained immunity; Innate immune system; MV130; Sublingual vaccine; Trained immunity-based vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Randomization will be done in a 1:1 ratio in blocks of 6, through a random list. It will be impossible for investigators to know to which group a subject will be assigned before being included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MV130 (Experimental): Suspension of 6 inactivated whole bacteria concentrates, that contains 90% of Gram positive bacteria (V104 S. pneumoniae 60%, V102 S. aureus 15%, V101 S. epidermidis 15%) and 10% of Gram negative bacteria (V113 K. pneumoniae 4%, V105 M. catarrhalis 3%, V103 H. influenzae 3%), at a concentration of 300 FTU/mL, equivalent to ~ 10^9 bacteria/mL.
  Interventions: Biological: MV130
- Placebo (Placebo Comparator): Sodium chloride 9 mg/mL and water for injection s.q. f 1 mL.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MV130 — Treatment administered sublingually
  Arms: MV130
Other: Placebo — Treatment administered sublingually
  Arms: Placebo

SUMMARY:
A mechanistic clinical trial with the aim to evaluate whether MV130 can induce the expression of a particular immune response (trained immunity) in peripheral blood cells. Therefore, the investigators are not evaluating efficacy in any disease or medical condition but rather assessing the immunological effect in immunogenicity of MV130 in healthy volunteers.

DETAILED DESCRIPTION:
Bacillus Calmette-Guérin (BCG) has been postulated as a strategy to prevent transmission and reduce the incidence of infectious diseases due to its ability to induce trained immunity. However, it is not recommended to vaccinate with live-attenuated vaccines, such as BCG, to certain vulnerable populations including immunocompromised patients. This issue can be overcome with inactivated preparations that mediate trained immunity such as MV130. The safety of MV130 in pilot studies in patients with immunodeficiency or solid organ recipients, has been highlighted in recent studies.

Based on the principles of trained immunity, it has recently been suggested that this concept can be further exploited in a next generation of anti-infectious vaccines: Trained immunity-based vaccines (TIbV). Thus, these vaccines may confer a broad protection far beyond to the nominal antigens they contain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that have provided written informed consent.
* Healthy males and females 18 to 65 years, both included, at the time of enrolment.
* Subjects who are able to provide cooperation and comply with dosing regimen.
* Women of childbearing age (from menarche) should submit a urine pregnancy test with a negative result at the time of enrolment in the trial.

Exclusion Criteria:

* Simultaneous participation in another clinical trial.
* Females who are pregnant or breast-feeding, or potential pregnant or breast-feeding females.
* Subjects who are allergic to any of the components included in MV130.
* Subjects with any concomitant disease or treatment that, according to the investigator criteria, may affect the development of this study, such as immunodeficiencies, malignancies involving bone marrow or lymphoid systems, medical treatment affecting the immune system (including corticosteroids, immunosuppressants, biological agents,…), human immunodeficiency virus, severe allergies, diabetes, hypertension, psychological disorders, etc.
* Subjects who have been vaccinated within 12 months before inclusion (flu or any other vaccine different from COVID-19 vaccine), or who have planned to be vaccinated during the clinical study (excluding the COVID-19 vaccine).
* Subjects who have had an infection that included fever and/or diarrhoea within 3 months before inclusion.
* Subjects under metformin treatment during the last month before inclusion in the clinical study or during the clinical trial*.
* Subjects under statins treatment during the last month before inclusion in the clinical trial or during*.

  *: these drugs interfere with metabolic pathways involved in trained immunity induction.
* Subjects who are allergic to any of the components included in the flu vaccine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Increase ex vivo in cytokine response | 70 days
  The primary outcome is the increase ex vivo in cytokine response (TNF-alfa, IL-6 and/or IL-1beta) in PBMCs upon secondary restimulation (MV130, lipopolysaccharide [LPS], inactivated Candida albicans, Resiquimod-R848, Poly I:C and/or phytohemagglutinin [PHA]) in MV130 vaccinated subjects compared to placebo group, at days 15, 45 and/or 70, with respect to baseline.

SECONDARY OUTCOMES:
Epigenetic and metabolic changes in purified monocytes from PBMCs, in a subgroup of MV130 vaccinated (n=12) versus placebo (n=12), at day 45 with respect to baseline. | 70 days
  It includes specific miRNA associated to trained immunity (miR155, miR146 and/or miR21, etc.) and histone marks (H3K4me3 and/or H3K27me3, among others), as epigenetic rewiring markers.
  It also includes lactate production, glucose consumption and mitochondrial activity as metabolic changes.
Changes in percentages of immune populations in peripheral blood including T and B cells, NK cells and subsets of monocytes, in MV130 group compared to placebo at days 15, 45 and/or 70, with respect to baseline. | 70 days
  Changes in percentages of immune populations in peripheral blood including T and B cells, NK cells and subsets of monocytes, in MV130 group compared to placebo at days 15, 45 and/or 70, with respect to baseline.
Change in MV130 non-specific response (T and B cells from PBMCs) in MV130 treated group compared to placebo. | 70 days
  It includes T cell proliferation (days 15, 45 and/or 70) by labelling T cells with carboxyfluorescein succinimidyl ester (CFSE) prior to restimulation with PHA, inactivated C. albicans and flu antigens. Also, change of cytokine production (such as IFN-gamma, IL-17 and/or IL-10) from T cells upon restimulation (LPS, inactivated Candida albicans, flu antigens and/or PHA) (days 15, 45 and/or 70 with respect to baseline).
  It also includes antibody production: cross-reactive serum IgG against viral components. Different viral proteins/peptides will be tested (days 45 and 70 with respect to baseline). Antibody responses against flu antigens (IgG and IgA in serum and IgA in saliva) will be evaluated (days 45 and 70 with respect to baseline).
MV130 specific response (T and B cells responses form PBMCs) in MV130 vaccinated group compared to placebo. | 70 days
  It includes T cell proliferation and cytokine production (IFN-gamma, IL-17 and/or IL-10) following restimulation with MV130 (days 15, 45 and/or 70 with respect to baseline).
  It also includes antibody production: MV130 specific IgG and IgA levels in serum and IgA levels in saliva (days 45 and/or 70 with respect to baseline). Individual bacteria contained in MV130 (i.e., S. pneumoniae) will be further tested for specific antibody production.
Change in baseline oral microbiota composition in MV130 treated group (days 45 and 70 with respect to baseline) compared to placebo, based on the 16S rRNA sequence phylogeny. | 70 days
  Change in baseline oral microbiota composition in MV130 treated group (days 45 and 70 with respect to baseline) compared to placebo, based on the 16S rRNA sequence phylogeny.
Rates of adverse events | 70 days
  The overall rate of adverse events in both groups
Classification of the Adverse events | 70 days
  Classification of the Adverse events during the trial
Rates of adverse reactions | 70 days
  The overall rate of adverse reactions in both groups
Classification of the Adverse reactions | 70 days
  Classification of the Adverse reactions during the trial
Percentage by type of adverse events | 70 days
  Percentage by type of adverse events occurred during the trial
Percentage of subject with adverse reactions | 70 days
  Percentage of subject experiencing adverse reactions during the trial
Timing of reaction appearance | 70 days
  Time from the first administration to appearance of the reaction
Classification of the adverse reaction according to the place of appearance | 70 days
  Classification of the adverse reaction in local or systemic, depending on the place of appearance

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Sánchez-Ramón, MD and PhD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clínico San Carlos, Madrid, Spain

REFERENCES:
- [Background] Netea MG, Dominguez-Andres J, Barreiro LB, Chavakis T, Divangahi M, Fuchs E, Joosten LAB, van der Meer JWM, Mhlanga MM, Mulder WJM, Riksen NP, Schlitzer A, Schultze JL, Stabell Benn C, Sun JC, Xavier RJ, Latz E. Defining trained immunity and its role in health and disease. Nat Rev Immunol. 2020 Jun;20(6):375-388. doi: 10.1038/s41577-020-0285-6. Epub 2020 Mar 4. PMID 32132681
- [Background] Sanchez-Ramon S, Conejero L, Netea MG, Sancho D, Palomares O, Subiza JL. Trained Immunity-Based Vaccines: A New Paradigm for the Development of Broad-Spectrum Anti-infectious Formulations. Front Immunol. 2018 Dec 17;9:2936. doi: 10.3389/fimmu.2018.02936. eCollection 2018. PMID 30619296
- [Background] Guevara-Hoyer K, Saz-Leal P, Diez-Rivero CM, Ochoa-Grullon J, Fernandez-Arquero M, Perez de Diego R, Sanchez-Ramon S. Trained Immunity Based-Vaccines as a Prophylactic Strategy in Common Variable Immunodeficiency. A Proof of Concept Study. Biomedicines. 2020 Jul 9;8(7):203. doi: 10.3390/biomedicines8070203. PMID 32660100
- [Background] Alecsandru D, Valor L, Sanchez-Ramon S, Gil J, Carbone J, Navarro J, Rodriguez J, Rodriguez-Sainz C, Fernandez-Cruz E. Sublingual therapeutic immunization with a polyvalent bacterial preparation in patients with recurrent respiratory infections: immunomodulatory effect on antigen-specific memory CD4+ T cells and impact on clinical outcome. Clin Exp Immunol. 2011 Apr;164(1):100-7. doi: 10.1111/j.1365-2249.2011.04320.x. PMID 21391984
- [Background] Garcia Gonzalez LA, Arrutia Diez F. Mucosal bacterial immunotherapy with MV130 highly reduces the need of tonsillectomy in adults with recurrent tonsillitis. Hum Vaccin Immunother. 2019;15(9):2150-2153. doi: 10.1080/21645515.2019.1581537. Epub 2019 Apr 17. PMID 30779677
- [Background] Nieto A, Mazon A, Nieto M, Calderon R, Calaforra S, Selva B, Uixera S, Palao MJ, Brandi P, Conejero L, Saz-Leal P, Fernandez-Perez C, Sancho D, Subiza JL, Casanovas M. Bacterial Mucosal Immunotherapy with MV130 Prevents Recurrent Wheezing in Children: A Randomized, Double-Blind, Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2021 Aug 15;204(4):462-472. doi: 10.1164/rccm.202003-0520OC. PMID 33705665
- [Background] Cirauqui C, Benito-Villalvilla C, Sanchez-Ramon S, Sirvent S, Diez-Rivero CM, Conejero L, Brandi P, Hernandez-Cillero L, Ochoa JL, Perez-Villamil B, Sancho D, Subiza JL, Palomares O. Human dendritic cells activated with MV130 induce Th1, Th17 and IL-10 responses via RIPK2 and MyD88 signalling pathways. Eur J Immunol. 2018 Jan;48(1):180-193. doi: 10.1002/eji.201747024. Epub 2017 Sep 14. PMID 28799230
- [Background] Vazquez A, Fernandez-Sevilla LM, Jimenez E, Perez-Cabrera D, Yanez R, Subiza JL, Varas A, Valencia J, Vicente A. Involvement of Mesenchymal Stem Cells in Oral Mucosal Bacterial Immunotherapy. Front Immunol. 2020 Nov 19;11:567391. doi: 10.3389/fimmu.2020.567391. eCollection 2020. PMID 33329530
- [Background] Del Fresno C, Garcia-Arriaza J, Martinez-Cano S, Heras-Murillo I, Jarit-Cabanillas A, Amores-Iniesta J, Brandi P, Dunphy G, Suay-Corredera C, Pricolo MR, Vicente N, Lopez-Perrote A, Cabezudo S, Gonzalez-Corpas A, Llorca O, Alegre-Cebollada J, Garaigorta U, Gastaminza P, Esteban M, Sancho D. The Bacterial Mucosal Immunotherapy MV130 Protects Against SARS-CoV-2 Infection and Improves COVID-19 Vaccines Immunogenicity. Front Immunol. 2021 Nov 18;12:748103. doi: 10.3389/fimmu.2021.748103. eCollection 2021. PMID 34867974
- [Background] Ochoa-Grullon J, Benavente Cuesta C, Gonzalez Fernandez A, Cordero Torres G, Perez Lopez C, Pena Cortijo A, Conejero Hall L, Mateo Morales M, Rodriguez de la Pena A, Diez-Rivero CM, Rodriguez de Frias E, Guevara-Hoyer K, Fernandez-Arquero M, Sanchez-Ramon S. Trained Immunity-Based Vaccine in B Cell Hematological Malignancies With Recurrent Infections: A New Therapeutic Approach. Front Immunol. 2021 Feb 12;11:611566. doi: 10.3389/fimmu.2020.611566. eCollection 2020. PMID 33679698
- [Background] Molero-Abraham M, Sanchez-Trincado JL, Gomez-Perosanz M, Torres-Gomez A, Subiza JL, Lafuente EM, Reche PA. Human Oral Epithelial Cells Impair Bacteria-Mediated Maturation of Dendritic Cells and Render T Cells Unresponsive to Stimulation. Front Immunol. 2019 Jun 28;10:1434. doi: 10.3389/fimmu.2019.01434. eCollection 2019. PMID 31316504